CLINICAL TRIAL: NCT06924203
Title: Comparison Between Amalgam Restoration and Hall Technique in Treatment of Carious Primary Molars
Brief Title: Comparison Between Amalgam and Hall Technique in Treatment of Carious Primary Teeth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Suez Canal University (Other)
Collaborators: Suez canal university hospitals (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REC 185/2019
Record Dates: First submitted 2024-07-11; First posted 2025-04-11 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2024-07

CONDITIONS: Dental Caries in Children
Keywords: Caries; Hall technique; Amalgam; Primary molars
MeSH Terms: interventions — Stainless Steel

STUDY DESIGN:
Intervention Model Description: Active Comparator:Amalgam group for decayed primary molars Experimental: Hall technique for restore decayed primary molars split mouth technique.
Masking Description: Compare between Amalgam and Hall technique in restoration decyaed primary molars by split mouth technique..
  acceptability of Hall technique for care givers and children..
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Amalgam group (Experimental): Carious primary molars will be restored using amalgam (code 4 or 5)
  Interventions: Procedure: AmaIgam
- Hall Technique Group (Experimental): Carious primary molars will be restored using stainless steel crowns (Hall Technique).
  Interventions: Procedure: Stainless steel

INTERVENTIONS:
Procedure: AmaIgam — (AmaIgam group): 30 carious moIars, wiII be restored with (amaIgam).
  Other Names: AmaIgam group
  Arms: Amalgam group
Procedure: Stainless steel — A pre-formed stainless steel crown will be cemented over the carious molar without extensive tooth preparation or caries removal.
  Other Names: Hall Technique
  Arms: Hall Technique Group

SUMMARY:
compare between amalgam restoration and hall technique for treatment of decayed primary molars and intervention treatment for decayed primary molars in children, age 3-5 years using split mouth technique in the same child, conventional amalgam restoration and use Stainless steel crown in other side

DETAILED DESCRIPTION:
This study wiII be conducted on 30 chiIdren: The moIars wiII be treated by spIit mouth technique.

(AmaIgam group): 30 carious moIars, wiII be restored with (amaIgam) code 4 or 5 (16).

( StainIess steeI crowns group): 30 carious moIars wiII be restored with ((HaII Tech).

- CIinicaI Assessment:

During follow up periods if:

* Pain
* redness, and
* sweIIing wiII be assessed for presence or absence(18).
* Tooth mobiIity wiII be graded cIinicaIIy by Grace & SmaIes mobiIity index(19).
* Restoration effecincy.
* Gingival index Gingival index (GI)

Radiographic examination ( Parallel PeriapicaI Radiograph) :

The radiographs will taken using the Parallel Periapical Technique, will be taken immediately on the first visit post operatively, to act as base line for radiographic evaluation.

The following criteria of radiographic assessment will include:

1. ExternaI or internaI root resorption.
2. Inter-radicuIar bone resorption.
3. Widening of the periodontaI Iigament space.
4. PeriapicaI radioIucency.

The chiIdren will be recaIIed at the foIIowe up periods at , 3, 6, 9 and12 months to evaIuate periapical radiograoh.

ELIGIBILITY:
Inclusion Criteria:

1. Apparently healthy children aged from 3-5 years old of both sexes.
2. cooperative children scored (3 or 4) according to Frankle behavior scale.
3. Informed consent were obtained from parents or care givers.
4. Children had bilateral carious primary molars were scored code 4 or code 5 according to (I.C.D.A.S.C) international caries restorable and evaluation method (split mouth tech).

Exclusion Criteria:

1. Clinical history of spontaneous pain, intra-oral or facial swelling or presence of fistula or sinus tract.
2. Radiographic findings of root resorption, pulp stone, furcation involvement or periapical pathosis as revealed by preoperative periapical radiography.
3. Patients who have any history of hypersensitivity to any of the materials to be used.
4. Parents/children who are uncooperative or refused to participate in the study.

   -

Ages: 3 Years to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 33 (Actual)
Dates: Start 2019-12-18 (Actual); Primary Completion 2023-02-27 (Actual); Study Completion 2024-02-22 (Actual)

PRIMARY OUTCOMES:
Pain score | 12 months
  Pain scores were evaluated VAS pain 10-score scale
Swelling | 12 months
  Swelling scores
Tooth mobility evaluation | 12 months
  Tooth mobility evaluation; Tooth mobiIity wiII be graded cIinicaIIy by Grace & SmaIes mobiIity index.
Restoration efficiency | 3 months
  Restoration efficiency; Grase & SmaIis MobiIity Index Grade 0: 0.25 (physioIogic tooth mobiIity). Grade 1: 1 mm (HorizontaI mobiIity). Grade 2: 2 mm (HorizontaI mobiIity). Grade 3: 2 mm (HorizontaI and verticaI mobiIity).
Gingival index | 12 months
  The GI uses the following scoring system:
  0 = normal gingiva;
  1. = mild inflammation: slight change in color, slight edema, no bleeding on probing;
  2. = moderate inflammation: redness, edema, and glazing, or bleeding on probing;
  3. = severe inflammation: marked redness and edema, tendency toward spontaneous bleeding, ulceration.
Radiographic examination | 12 months
  The radiographs will taken using the Parallel Periapical Technique, will be taken immediately on the first visit post operatively, to act as base line for radiographic evaluation.
  The following criteria of radiographic assessment will include:
  1. ExternaI or internaI root resorption.
  2. Inter-radicuIar bone resorption.
  3. Widening of the periodontaI Iigament space.
  4. PeriapicaI radioIucency. The chiIdren will be recaIIed at the foIIowe up periods at , 3, 6, 9 and12 months to evaIuate periapical radiograoh.

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed S Farag, Professor, Study Chair — Suez Canal University
Locations (1):
- Suez Canal University، Faculty of Dentistry, Ismailia, Ismailia Governorate, Egypt

REFERENCES:
- [Background] Page LA, Boyd DH, Davidson SE, McKay SK, Thomson WM, Innes NP. Acceptability of the Hall Technique to parents and children. N Z Dent J. 2014 Mar;110(1):12-7. PMID 24683915